CLINICAL TRIAL: NCT01395277
Title: Effects of Dietary Flavanols on Cutaneous, Peripheral, and Cerebral Vascular Function in Young and Old Humans
Brief Title: Role of Flavanols In Cardiovascular Function in Healthy Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Robert M. Brothers, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011-05-0029
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Aging
Keywords: Nitric Oxide; Vascular Function; Aging; Blood Pressure; Arterial Stiffness; Cardiovascular Disease; Cerebral Blood Flow
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Flavanol first then Low Flavanol (Experimental): The measurements will be made on all study participants on two separate occasions; 1) before and 2 hours following consumption of a beverage with "high" flavanol content and 2) before and 2 hours following consumption of a beverage with "low" flavanol content.
  Interventions: Dietary Supplement: High Flavanol first then Low Flavanol
- Low Flavanol first then High Flavanol (Experimental): The measurements will be made on all study participants on two separate occasions; 1) before and 2 hours following consumption of a beverage with "low" flavanol content and 2) before and 2 hours following consumption of a beverage with "high" flavanol content.
  Interventions: Dietary Supplement: Low Flavanol first then High Flavanol

INTERVENTIONS:
Dietary Supplement: High Flavanol first then Low Flavanol — The high flavanol trial will be performed following consumption of a beverage containing 1,050 mg of commercially available Cocoa Flavanols which will be mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption. The low flavanol trial will be performed following consumption of a beverage containing 0 mg of Cocoa Flavanols which will be mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption.
  Other Names: dark chocolate beverage
  Arms: High Flavanol first then Low Flavanol
Dietary Supplement: Low Flavanol first then High Flavanol — The low flavanol trial will be performed following consumption of a beverage containing 0 mg of Cocoa Flavanols which will be mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption. The high flavanol trial will be performed following consumption of a beverage containing 1,050 mg of commercially available Cocoa Flavanols which will be mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption.
  Other Names: chocolate; Mars Incorporated
  Arms: Low Flavanol first then High Flavanol

SUMMARY:
Groups of naturally occurring compounds called flavonoids are found in foods such as fruits and vegetables, red wine, tea, dark chocolate and cocoa products. Diets rich in flavonoids are associated with decreased risk for cardiovascular disease and major cardiovascular events (i.e. myocardial infarction) and have been shown to improve blood pressure, insulin sensitivity, and vascular function in a variety populations (Type II diabetes, elderly, smokers, etc.). The presumed beneficial effects of these compounds are thought to act through their inherent ability to scavenge free radicals. Specifically flavonoids scavenge superoxide anions which are free radicals that react with nitric oxide (NO) to produce peroxynitrite. The formation of peroxynitrite ultimately reduces the bioavailability of NO which is essential for vasodilation and thus vascular health and function. Normal aging is associated with impaired endothelial function, which presumably is due to less than optimal levels of NO bioavailability. Therefore, interventions that can increase NO bioavailability would be expected to improve microvascular function and vascular health in this population. The purpose of this study is to investigate the effects of dietary flavonoid supplementation on the vasodilatory capacity of the cutaneous vasculature, as well as on cerebral vascular reactivity and arterial stiffness in young and old humans. This study will test the hypothesis that acute dietary flavonoid treatment will improve impaired cutaneous vasodilatory capacity, cerebral vasomotor reactivity, and reduce arterial stiffness in older but not young humans.

DETAILED DESCRIPTION:
Role of nitric oxide in vascular function. Nitric oxide (NO) is an important signaling molecule involved in many physiological processes. Of particular interest is its role in endothelial function and blood flow regulation. In response to heat or sheer stress against the walls of blood vessels, the endothelial layer of blood vessels releases NO, which causes smooth muscle in the vessel wall to relax and the vessel to dilate. Environmental heat-stress leads to an increase in skin blood flow to allow for improved heat loss from the body surface to the environment, and relies on NO. Normal aging reduces NO bioavailability leading to an impaired ability to increase skin blood flow in response to environmental heat-stress. Additionally, cerebral blood flow is reduced and arterial stiffness is increased in the normal aging process which is at least partially attributed to reductions in NO bioavailability.

Effects of dietary flavonoids. As previously mentioned Flavonoids are a group of natural compounds found in vegetables, fruits, wine, tea, and cocoa. Flavanols are a subfamily of flavonoids, and are quantitatively the most important compound in flavonoid family in western diets. Flavanol intake has been shown to improve vascular health, as well as increase insulin sensitivity, decrease blood pressure, reduce platelet aggregation, and enhance cerebral blood flow. The basic chemical features of flavanol allows them to act as classic antioxidants to scavenge free-radicals decreasing oxidant level in cells. High levels of free radicals, especially superoxide, can reduce the bioavailability of NO and thus any NO-mediated actions. Cocoa and cocoa products are potent sources of flavanols, and therefore have been used extensively as a dietary intervention to study the effects of flavanol supplementation on various disease states.

Impairments in vascular health in the normal aging process. The ability to increase skin blood flow in response to environmental heat-stress is lost with normal aging, especially when individuals exceed 65 years of age. An attenuated skin blood flow response during exposure to environmental heat stress would place these older individuals at an increased risk for heat-related illness or death. The ability to raise skin blood flow with rising skin temperature has been demonstrated to have a large nitric oxide component, so a deficit in NO bioavailability, which is also consistently observed in aging populations, could presumably lead to the attenuated skin blood flow response to heat stress. Furthermore, it is well documented that cerebral blood flow is reduced while arterial stiffness is increased in the normal aging process. In regard to the reduction in NO in aging populations, flavanol supplementation has been shown to decrease production of free radicals, which can scavenge and reduce NO levels thereby improving indices of vascular health including flow mediated vasodilation. Therefore, flavanol supplementation may maintain NO bioavailability at optimal levels, and provide a feasible way for aging populations to maintain vascular health and prevent heat-related illness and death.

Significance:

This study will address the mechanisms of impaired cutaneous and cerebral blood flow as well as increased arterial stiffness that can occur in aging populations. Furthermore, if the hypothesis is correct, findings from this study will provide evidence for the efficacy of flavanols to be used (as a simple and safe lifestyle intervention) to reverse or combat impaired vascular function that commonly occurs in older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between 18 - 26 years old
* Males and Females between 65 - 80 years old

Exclusion Criteria:

* cardiovascular disease
* metabolic disease
* neurological disease
* Pregnant lady
* Current smoker (or regularly smoked within last year)
* Currently taking medications known to effect the autonomic nervous system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Matthew Brothers, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin: Environmental and Autonomic Physiolgy Laboratory, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Flavanol First Then Low Flavanol: The measurements will be made on all study participants on two separate visits to the laboratory; On the first visit measurements will be made before (baseline) and 2 hrs post consumption of a beverage with "high" flavanol content. On the second study visit measurements will be made before and 2 hrs following consumption of a beverage with "low" flavanol content.
  During the first visit the high flavanol measures will be performed before and 2 hours following consumption of a beverage containing 1,050 mg of Cocoa Flavanols mixed into 250 ml of distilled water. Measurements will be performed 2 hrs after consumption. During the second visit the low flavanol measures will be performed following consumption of a beverage containing 0 mg of Cocoa Flavanols mixed into 250 ml of distilled water. Measurements will be performed 2 hrs after consumption.
- Low Flavanol First Then High Flavanol: The measurements will be made on all study participants on two separate visits to the laboratory; On the first visit measurements will be made before (baseline) and 2 hrs post consumption of a beverage with "low" flavanol content. On the second study visit measurements will be made before and 2 hrs following consumption of a beverage with "high" flavanol content.
  During the first visit the low flavanol measures will be performed before and 2 hours following consumption of a beverage containing 0 mg of Cocoa Flavanols mixed into 250 ml of distilled water. Measurements will be performed 2 hrs after consumption. During the second visit the high flavanol measures will be performed following consumption of a beverage containing 1,050 mg of Cocoa Flavanols mixed into 250 ml of distilled water. Measurements will be performed 2 hrs after consumption.
Period: Overall Study
Arm/Group | High Flavanol First Then Low Flavanol | Low Flavanol First Then High Flavanol
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 15 young and 15 elderly subjects participated in portion of the protocol
Groups:
- High Flavanol First Then Low Flavanol: The measurements will be made on all study participants on two separate visits to the laboratory; On the first visit measurements will be made before (baseline) and 2 hrs post consumption of a beverage with "high" flavanol content . On the second study visit measurements will be made before and 2 hrs following consumption of a beverage with "low" flavanol content.
  During the first visit the high flavanol measures will be performed following consumption of a beverage containing 1,050 mg of Cocoa Flavanols mixed into 250 ml of distilled water. Measurements will be performed 2 hrs after consumption. During the second visit the placebo trial (low flavanol group) will be performed following consumption of a beverage containing 0 mg of Cocoa Flavanols mixed into 250 ml of distilled water. Measurements will be performed 2 hrs after consumption.
- Low Flavanol First Then High Flavanol: The measurements will be made on all study participants on two separate visits to the laboratory; On the first visit measurements will be made before (baseline) and 2 hrs post consumption of a beverage with "low" flavanol content. On the second study visit measurements will be made before and 2 hrs following consumption of a beverage with "high" flavanol content.
  During the first visit the low flavanol measures will be performed following consumption of a beverage containing 0 mg of Cocoa Flavanols mixed into 250 ml of distilled water. Measurements will be performed 2 hrs after consumption. During the second visit the high flavanol measures will be performed following consumption of a beverage containing 1,050 mg of Cocoa Flavanols mixed into 250 ml of distilled water. Measurements will be performed 2 hrs after consumption.
- Total: Total of all reporting groups
Arm/Group | High Flavanol First Then Low Flavanol | Low Flavanol First Then High Flavanol | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (2.8) | 67.5 (2.9) | 68.0 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Mean Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 85 (8) | 88 (7) | 87 (6)

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Blood Flow Response to Local Heating of the Skin.
Description: Local heating of the cutaneous vasculature to 42 degree C is commonly used to evoke a maximal skin blood flow response (only at the site of local heating). This response is almost entirely dependent on nitric oxide mediated vasodilation.
Time Frame: prior to (baseline) and 2 hours post beverage consumption
Measure: Mean (Standard Deviation); unit: percent change in mean skin blood flow
Groups:
- High Flavanol: The measurements will be made on all study participants on two separate occasions; 1) before and 2 hours following consumption of a beverage with "high" flavanol content (experimental trial), and 2) before and 2 hours following consumption of a beverage with "low" flavanol content (placebo trial).
  CocoaVia Dark Chocolate Flavored Drink: The experimental trial (high flavanol group) will be performed following consumption of a beverage containing 1,050 mg of Cocoa Flavanols. This cocoa flavanol powder will be purchased from Mars Incorporated (Hackettstown, New Jersey) and will be mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption.
- Low Flavanol: The measurements will be made on all study participants on two separate occasions; 1) before and 2 hours following consumption of a beverage with "high" flavanol content (experimental trial), and 2) before and 2 hours following consumption of a beverage with "low" flavanol content (placebo trial).
  Placebo Trial: CocoaVia Dark Chocolate Flavored Drink: The placebo trial (low flavanol content) will be performed following consumption of a beverage containing 75 mg of Cocoa Flavanols. This cocoa flavanol powder will be purchased from Mars Incorporated (Hackettstown, New Jersey) and will be mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption.
Arm/Group | High Flavanol | Low Flavanol
Number analyzed (Participants) | 30 | 30
percent change in mean skin blood flow | 68 (10.6) | 70 (12.3)

2. Secondary Outcome: Pulse Wave Velocity / Arterial Stiffness
Description: Assessment of pulse wave velocity in the common carotid artery and the femoral artery provides an index of arterial stiffness.
Time Frame: Prior to (baseline) and 2 hours following beverage consumption
Measure: Mean (Standard Deviation); unit: cm / sec
Groups:
- High Flavanol: The measurements will be made on all study participants on two separate occasions; 1) before and 2 hours following consumption of a beverage with "high" flavanol content, and 2) before and 2 hours following consumption of a beverage with "low" flavanol content.
  The high flavanol measures will be performed following consumption of a beverage containing 1,050 mg of Cocoa Flavanols mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption. The low flavanol measures will be performed following consumption of a beverage containing 0 mg of Cocoa Flavanols mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption.
- Low Flavanol: The measurements will be made on all study participants on two separate occasions; 1) before and 2 hours following consumption of a beverage with "low" flavanol content, and 2) before and 2 hours following consumption of a beverage with "high" flavanol content.
  The low flavanol measures will be performed following consumption of a beverage containing 0 mg of Cocoa Flavanols mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption. The hihg flavanol measures will be performed following consumption of a beverage containing 1,0500 mg of Cocoa Flavanols mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption.
Arm/Group | High Flavanol | Low Flavanol
Number analyzed (Participants) | 30 | 30
cm / sec | 2.5 (0.2) | 2.7 (.30)

ADVERSE EVENTS:
Time Frame: 4 years, 2 months
Description: No adverse events occurred
Groups:
- High Flavanol First Then Low Flavanol: The measurements will be made on all study participants on two separate occasions; 1) before and 2 hours following consumption of a beverage with "high" flavanol content, and 2) before and 2 hours following consumption of a beverage with "low" flavanol content.
  The high flavanol measures will be performed following consumption of a beverage containing 1,050 mg of Cocoa Flavanols mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption. The low flavanol measures will be performed following consumption of a beverage containing 0 mg of Cocoa Flavanols mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption.
- Low Flavanol First Then High Flavanol: The measurements will be made on all study participants on two separate occasions; 1) before and 2 hours following consumption of a beverage with "low" flavanol content, and 2) before and 2 hours following consumption of a beverage with "high" flavanol content.
  The low flavanol measures will be performed following consumption of a beverage containing 0 mg of Cocoa Flavanols mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption. The high flavanol measures will be performed following consumption of a beverage containing 1,050 mg of Cocoa Flavanols mixed into 250 ml of distilled water. The subjects will consume this beverage and measurements will be performed 2 hours after consumption.
Arm/Group | High Flavanol First Then Low Flavanol | Low Flavanol First Then High Flavanol
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No